CLINICAL TRIAL: NCT06426927
Title: A Colorectal Cancer Educational Intervention in the Latino Community Assessing the Feasibility of Recruitment & Retention Via a Church-Based Approach: Identification of Novel Barriers to Cancer Clinical Trial Enrollment
Brief Title: PeLear CCC: Proyecto Latino Contra Cancer Colorrectal
Acronym: PeLear CCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-2980; CTSC0205 (Other Grant/Funding Number: NCTraCS Institute)
Record Dates: First submitted 2024-05-08; First posted 2024-05-23 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Rectal Cancer; Colon Cancer; Colon Rectal Cancer; Rectal Neoplasms; Colon Adenocarcinoma; Hereditary Nonpolyposis Colon Cancer
Keywords: Colorectal Cancer; Latino; Barriers; Cancer Clinical Trials; Spanish; Familial Colorectal Cancer; Lynch Syndrome; Hispanic
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Videos (Experimental): Enrolled participants will watch three educational videos in Spanish pertaining to: (1) Colorectal Cancer (CRC) symptoms; (2) CRC risk factors and (3) CRC facts, screening, treatment, and Cancer Clinical Trials (CCT).
  Interventions: Other: Colorectal Cancer Educational Videos in Spanish

INTERVENTIONS:
Other: Colorectal Cancer Educational Videos in Spanish — Enrolled participants will watch three educational videos on Colorectal Cancer (CRC) in Spanish. Knowledge on CRC symptoms, risk factors, facts, screening and treatment will be assessed before and immediately after the educational video and at 30 +/- 7 days. In addition, the association between increase in CRC knowledge and willingness to participate in Cancer Clinical Trials (CCT) will be explored.

SUMMARY:
The study aims to recruit 60 Spanish speaking individuals who identify as Latinos, are 18 years or older and attend the Saint Thomas More (STM) Church in Chapel Hill. Study participants will be asked to attend an educational session at STM Church during which their baseline knowledge on colorectal cancer (CRC) and willingness to participate in cancer clinical trials (CCT) will be assessed through a questionnaire in Spanish. Following this, participants will watch three educational videos on CRC in Spanish. After watching the videos, CRC knowledge and willingness to participate in CCTs will be reassessed. Thirty +/- 7 days after participation in the educational session, participants will be invited back at STM Church in order to complete a follow-up questionnaire assessing CRC knowledge, willingness to participate in CCTs and perceived barriers preventing Latinos from participating in CCTs. Twenty of the 60 recruited participants will be asked to participate in a qualitative one-on-one interview aimed at identifying barriers preventing Latinos from participating in CCTs.

It should be noted that cancer is the leading cause of death in the United States (US) Latino community, with CRC accounting for 10% of this overall mortality. Despite this, Latinos suffer from disparities in access to care, cancer screening, treatment, and representation in CCTs. In fact, although Latino individuals are among the largest and fastest growing communities of color in the US, currently comprising 18.7%, their representation in CCTs remains low. This is of concern because: 1) advances arising from trials with limited Latino representation may not be applicable to the Latino population, and 2) decreased Latino participation in CCTs may delay Latino access to novel therapies in a timely fashion. The investigators conducting this study believe that low cancer-specific health knowledge may be impacting Latino representation and willingness to participate in CCTs and can be addressed through culturally and linguistically appropriate community-based educational interventions. Latino CCT underrepresentation is a multifaceted phenomenon and bidirectional barriers at the physician-, healthcare system-, and patient-level are significant contributors. Therefore, understanding the multiple driving forces and barriers is essential to identifying potential targets for improvement.

DETAILED DESCRIPTION:
This pilot project aims to address the Clinical and Translational Science (CTS) roadblock of underrepresentation of Latinos in cancer clinical trials (CCTs) through a community-based, culturally, and linguistically appropriate educational intervention aimed at increasing health knowledge on a specific cancer. Colorectal cancer (CRC) will be the "use case" and the church will be the venue for Latino recruitment. This project will lead to the identification of novel Latino-perceived barriers to CCT enrollment, which will be applicable in other fields of medicine aiming to increase Latino CCT enrollment. The investigators believe that one barrier to recruitment for CCTs is low health education, specifically regarding cancers affecting the community, such as CRC, a commonly diagnosed cancer in the US Latino population. Therefore, the hypothesis that an increase in health knowledge in Latinos on a specific cancer mediates a change in their willingness to participate in CCTs will be tested. To do this, three educational CRC videos in Spanish will be created. The first video will review CRC symptoms, the second video will review CRC risk factors while the third video will provide information on CRC facts, screening, treatment and CCTs. In addition, a translated, non-validated questionnaire based on 3 sub-scales from 2 CRC knowledge questionnaires previously validated in English will be developed and pilot tested. Therefore, the Specific Aims of this Pilot Project are to:

1. Identify novel Latino-perceived barriers to participation in CCTs.
2. Assess the association between an educational video and CRC knowledge.
3. Assess the potential relationship between an increase in health knowledge of a specific cancer via an educational video in Spanish and willingness to participate in CCTs.

To achieve these aims, recruit 60 Latino, Spanish speaking attendees of the Saint Thomas More (STM) Church in Chapel Hill will be recruited. The study will consist of three Study Days:

1. Study Day 1: Enrolled participants will be asked to attend an educational session at STM Church. During the educational session their baseline knowledge on CRC and their baseline willingness to participate in CCTs will be assessed through a questionnaire in Spanish. Following this, participants will watch three educational CRC videos in Spanish and then their CRC knowledge as well as their willingness to participate in CCTs will be reassessed.
2. Study Day 2: Thirty +/- 7 days after the educational session, participants will be asked to return to STM Church in order to complete a follow-up questionnaire in Spanish. The questionnaire will assess their level of retainment of CRC knowledge, their willingness to participate in CCTs as well as assess in an open-ended fashion their perceived barriers to CCT participation.
3. Study Day 3: Twenty of the 60 enrolled participants will be asked to participate in a qualitative one-on-one interview aimed at identifying Latino perceived barriers to CCT participation.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking
* Identifying as Latino
* 18 years or older

Exclusion Criteria:

* Non-Spanish speakers
* Not identifying as Latino
* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José G. Guillem, MD, MPH, MBA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Saint Thomas More Church, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sepucha KR, Feibelmann S, Cosenza C, Levin CA, Pignone M. Development and evaluation of a new survey instrument to measure the quality of colorectal cancer screening decisions. BMC Med Inform Decis Mak. 2014 Aug 20;14:72. doi: 10.1186/1472-6947-14-72. PMID 25138444
- [Background] American Cancer Society. Cancer Facts & Figures for Hispanic/Latino People 2021-2023. Atlanta: American Cancer Society, Inc. 2021.
- [Background] Power E, Simon A, Juszczyk D, Hiom S, Wardle J. Assessing awareness of colorectal cancer symptoms: measure development and results from a population survey in the UK. BMC Cancer. 2011 Aug 23;11:366. doi: 10.1186/1471-2407-11-366. PMID 21859500
- See also: Bowel Cancer Awareness Measure — https://www.cancerresearchuk.org/sites/default/files/health_professional_bowel_cam_toolkit_version_2.1_09.02.11.pdf
- See also: Racial and Ethnic Composition of the United States — https://www.census.gov/library/stories/2021/08/improved-race-ethnicity-measures-reveal-united-states-population-much-more-multiracial.html
- See also: National Cancer Institute Triennial Inclusion of Women and Minorities in Clinical Research Report — https://report.nih.gov/sites/report/files/docs/NCITriennialInclusionReportFY2019_FY2021Final.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Videos
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Educational Videos
Number analyzed (Participants) | 60
Age, Continuous [Mean (Full Range); unit: years] | 51.3 [20 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 1
  Unknown or Not Reported | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Attitudes Regarding Participation in Clinical Trials-Conceptual Themes (General Clinical Trials)
Description: Twenty participants were invited for qualitative interviews. Qualitative, semi-structured, one-on-one interviews will be performed in Spanish. The interviews will be recorded and transcribed. The ATLAS.ti software will be used for the transcript analysis. The top 2 conceptual themes for attitudes regarding general clinical trials will be reported in terms of percentage of participants.
Time Frame: 30 days after participation in Study Day 2
Population: Per the protocol, a traditional "power analysis" is not directly applicable to the qualitative, semi-structured one-on-one interview aspect of the trial. Based on published methodologies to assess the adequate sample to reach "saturation", 20 participants were invited for qualitative interviews.
Measure: Number; unit: percentage of participants
Arm/Group | Educational Videos
Number analyzed (Participants) | 20
percentage of participants
  Work is a priority | 85
  Preference for communicating in Spanish | 80

2. Primary Outcome: Attitudes Regarding Participation in Cancer Clinical Trials-Conceptual Themes (Cancer Clinical Trials)
Description: Twenty participants were invited for qualitative interviews. Qualitative, semi-structured, one-on-one interviews will be performed in Spanish. The interviews will be recorded and transcribed. The ATLAS.ti software will be used for the transcript analysis. The top 2 conceptual themes for attitudes regarding cancer clinical trials will be reported in terms of percentage of participants.
Time Frame: 30 days after participation in Study Day 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Educational Videos
Number analyzed (Participants) | 20
percentage of participants
  Fear of side effects | 60
  Knowledge is "peace of mind" | 45

3. Primary Outcome: Perceptions of Latino Community for Increasing Enrollment in Randomized Clinical Trials-Conceptual Themes (General Clinical Trials)
Description: Twenty participants were invited for qualitative interviews. Qualitative, semi-structured, one-on-one interviews will be performed in Spanish. The interviews will be recorded and transcribed. The ATLAS.ti software will be used for the transcript analysis. The top 2 conceptual themes for perceptions of the Hispanic/Latino community will be reported in terms of percentage of participants.
Time Frame: 30 days after participation in Study Day 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Educational Videos
Number analyzed (Participants) | 20
percentage of participants
  Go to where Latinos congregate | 90
  Video-based communication is preferred | 80

4. Primary Outcome: Holistic Themes
Description: Twenty participants were invited for qualitative interviews. Qualitative, semi-structured, one-on-one interviews will be performed in Spanish. The interviews will be recorded and transcribed. The ATLAS.ti software will be used for the transcript analysis. The top 3 holistic themes will be reported in terms of percentage of participants.
Time Frame: 30 days after participation in Study Day 2
Measure: Number; unit: percentage of participants
Arm/Group | Educational Videos
Number analyzed (Participants) | 20
percentage of participants
  Perception of Clinical Trials (CTs): "Positives Outweigh the Negatives" | 58
  Attitudes regarding CTs: "Factors Alleviating/ Exacerbating Fear Influence Attitude" | 100
  Attitudes regarding Cancer CTs: "Peace of Mind vs. Bodily Invasion/Side Effects Influence Attitude" | 45

5. Secondary Outcome: Association of Educational Videos on Knowledge of Colorectal Cancer Symptoms
Description: Use of appropriate statistical measures to compare total number of correct responses across three time points (at baseline, post-video and 30+/- 7 days follow-up) accounting for multiple observations within subjects. Knowledge pertaining to Colorectal Cancer (CRC) symptoms will be assessed using the "Knowledge of Warning Signs" questions from the "Bowel Cancer Awareness Measure". Potential answers include "Yes", "No" and "Don't Know". The overall score will range from 0 to 9 and it is anticipated that average scores will increase after the intervention. Higher scores imply greater knowledge of symptoms.
Time Frame: On Study Day 1: Immediately before (baseline) and immediately post-video (within 30 minutes); Study Day 2: 30 +/- 7 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Educational Videos
Number analyzed (Participants) | 60
score on a scale
  Study Day 1: Baseline | 4.10 (0.36)
  Study Day 1: Post-video | 7.23 (0.32)
  Study Day 2: 30 +/- 7 days | 6.95 (0.29)
Statistical Analysis 1: Comparison: Educational Videos; Post-video vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Educational Videos; Study Day 2: 30 +/- 7 days vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA

6. Secondary Outcome: Association of Educational Videos on Knowledge of Colorectal Cancer Risk Factors
Description: Use of appropriate statistical measures to compare mean of correct responses across three time points (at baseline, post-video and 30+/- 7 days follow-up) accounting for multiple observations within subjects. Knowledge pertaining to Colorectal Cancer (CRC) risk factors will be assessed using the "Knowledge of Risk Factors" questions from the "Bowel Cancer Awareness Measure". This scale is measured using a Likert 1-5 scale with "1" corresponding to "Strongly Disagree" and "5" corresponding to "Strongly Agree". The overall score will range from 1 to 5 and it is anticipated that the average scores will increase after the intervention. Higher scores imply greater knowledge of risk factors.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Educational Videos
Number analyzed (Participants) | 60
score on a scale
  Study Day 1: Baseline | 3.06 (0.08)
  Study Day 1: Post-video | 4.08 (0.15)
  Study Day 2: 30 +/- 7 days | 3.93 (0.12)
Statistical Analysis 1: Comparison: Educational Videos; Post-video vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Educational Videos; Study Day 2: 30 +/- 7 days vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA

7. Secondary Outcome: Association of Educational Videos on Knowledge of Colorectal Cancer Screening and Facts
Description: Use of appropriate statistical measures to compare mean of correct responses across three time points (at baseline, post-video and 30+/- 7 days follow-up) accounting for multiple observations within subjects. Knowledge of Colorectal Cancer (CRC) screening and general facts will be assessed using nine questions from the "Colorectal Cancer Screening Decision Quality Instrument (CRC-DQI)". The overall score will range from 0 to 9 and it is anticipated that average scores will increase after the intervention. Higher scores imply greater knowledge of colorectal cancer screening and facts.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Educational Videos
Number analyzed (Participants) | 60
score on a scale
  Study Day 1: Baseline | 3.80 (0.20)
  Study Day 1: Post-video | 6.05 (0.20)
  Study Day 2: 30 +/- 7 days | 5.12 (0.22)
Statistical Analysis 1: Comparison: Educational Videos; Post-video vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Educational Videos; Study Day 2: 30 +/- 7 days vs. Baseline; Test type: Superiority; p < 0.0001, ANOVA

8. Secondary Outcome: Association of Watching the Video and Willingness to Participate in Cancer Clinical Trials
Description: Appropriate statistical measures on the paired responses of participants will be used to test the association between watching the video and willingness to participate in CCTs. The mediating effect of Study Day 1 post-video health knowledge levels (M) on the relationship between educational video (X) and willingness to participate in CCTs (Y) will be explored. In a structural equation model with a series of mixed-effects generalized linear models, Y will be predicted by both X and M, combining the estimated relationship of M and Y. The mediated indirect effect (from X to Y, through M) will then be estimated and tested using the bootstrapping method with 1,000 replications, and the proportion of the effect being mediated will be reported as the effect size. The number of participants who responded "Yes" to willingness to participate in cancer clinical trials are reported in the data table.
Time Frame: On Study Day 1: Immediately before (baseline) and immediately post-video (within 30 minutes) after the video projection
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Videos
Number analyzed (Participants) | 60
Participants
  Study Day 1: Baseline | 55
  Study Day 1: Post-video | 54
Statistical Analysis 1: Comparison: Educational Videos; Pre-video to post video, without covariates; Test type: Superiority; p = 0.56, Mixed Models Analysis; Average Causal Mediated Effect (ACME) = 0.01

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored from the time of signing informed consent through study completion, up to 30 days for participants involved in the educational video only and up to 60 days for those who participated in the qualitative interviews.
Description: The participants in the study completed questionnaires pre- and post- an educational video. The risks associated with this study were minimal and the participants were not at risk for mortality or serious adverse events as a function of participating in this study. Because this study investigated the impact of an educational intervention, All-Cause Mortality and Serious Adverse events were not monitored or assessed.
Arm/Group | Educational Videos
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT06426927/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT06426927/ICF_001.pdf